CLINICAL TRIAL: NCT06478602
Title: Implications of Fecal Microbiota Transplantation in Modulating the Effects of Liver Cirrhosis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cristian Ichim (Other)
Responsible Party: Sponsor-Investigator, Cristian Ichim, Principal Investigator, Academic Emergency County Hospital Sibiu
Organization: Academic Emergency County Hospital Sibiu (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: No: 3505/15.02.2023
Record Dates: First submitted 2024-06-23; First posted 2024-06-27 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — Fecal Microbiota Transplantation; Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fecal microbiota transplantation (FMT) in patients with liver cirrhosis (Experimental): The experimantal group will receive fecal transplantation from a healthy donor. The study results will be obtained from analyzing the progression observed in imaging and laboratory tests (blood and fecal matter) as well as the patients clinical condition - compared to the initial phase and the control group. Patients will undergo fecal transplantation using a minimum of 70 grams of material collected and tested from a healthy donor. The fecal matter will be transferred into the cecum using a colonoscope.
  Interventions: Biological: Fecal microbiota transplantation
- Control (No Intervention): The control group will include patients who will be monitored for their progress while receiving standard treatment.

INTERVENTIONS:
Biological: Fecal microbiota transplantation — Performing a colonoscopy with fecal microbiota transplantation at the level of the cecum.
  Other Names: Colonoscopy
  Arms: Fecal microbiota transplantation (FMT) in patients with liver cirrhosis

SUMMARY:
The study aims to investigate the beneficial effects of fecal transplantation in patients diagnosed with liver cirrhosis (regardless of etiology).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of liver cirrhosis according to current protocols.
* Conscious and cooperative adult patients.

Exclusion Criteria:

* Patients with hemodynamic and/or respiratory instability.
* Patients with contraindications for colonoscopy or fecal transplantation.
* Patients with acute or chronic infections with HIV, Tuberculosis, MDR Enterobacteria, CMV, parasites, fungi.
* Associated oncological pathology.
* Patients with other causes of severe immunodeficiencies.
* Lack of compliance with the conditions imposed by the research project.
* Patients who do not sign the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Implications of fecal microbiota transplantation in modulating the effects of liver cirrhosis. | Up to 3 months
  The transfer of microbiota could potentially influence hepatic fibrosis via the gut-liver axis, as well as other complications caused by cirrhosis such as encephalopathy, ascites etc.
Implications of fecal microbiota transplantation in modulating the condition of other organs. | Up to 3 months
  The transfer of microbiota could potentially modulate the function of other major organs in the body.

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Birlutiu, Prof. Dr., Study Chair — County Clinical Emergency Hospital of Sibiu; Adrian Boicean, Prof. Dr., Study Director — County Clinical Emergency Hospital of Sibiu
Locations (1):
- County Clinical Emergency Hospital of Sibiu, Sibiu, Romania

IPD SHARING:
Plan to Share IPD: No
The study results will be made public and other researchers will be able to receive the anonymized database upon reasonable request.

REFERENCES:
- [Background] Boicean A, Birlutiu V, Ichim C, Brusnic O, Onisor DM. Fecal Microbiota Transplantation in Liver Cirrhosis. Biomedicines. 2023 Oct 30;11(11):2930. doi: 10.3390/biomedicines11112930. PMID 38001930
- [Background] Boicean A, Ichim C, Todor SB, Anderco P, Popa ML. The Importance of Microbiota and Fecal Microbiota Transplantation in Pancreatic Disorders. Diagnostics (Basel). 2024 Apr 23;14(9):861. doi: 10.3390/diagnostics14090861. PMID 38732276
- [Background] Boicean A, Birlutiu V, Ichim C, Anderco P, Birsan S. Fecal Microbiota Transplantation in Inflammatory Bowel Disease. Biomedicines. 2023 Mar 27;11(4):1016. doi: 10.3390/biomedicines11041016. PMID 37189634